CLINICAL TRIAL: NCT06802237
Title: Clinical Method Development and Standardization Plan for Measuring Hair Growth
Brief Title: Development and Standardization Methods
Status: Completed | Type: Observational
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: NB240033-NB-V
Record Dates: First submitted 2025-01-23; First posted 2025-01-31 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — Assess and Evaluate hair growth and scalp health

SUMMARY:
The objective of this study is to establish a standardized methodology that integrates various parameters to comprehensively assess and evaluate hair growth and scalp health.

DETAILED DESCRIPTION:
A total of 25 participants, consisting of 13 males and 12 females who have complaints of androgenetic alopecia (AGA) will be enrolled.

This research seeks to develop and implement a robust and standardized approach that incorporates a diverse range of parameters. These parameters include:

* Measurement of hair regrowth from AGA-affected area.
* Number of new hairs from the AGA-affected area and tattoo area.
* Evaluation of hair strength through tensile testing.
* Assessment of hair length
* Global picture of head crown
* Quantitative analysis of scalp keratin levels.
* Visual documentation and quantitative scoring of baldness using the Norwood-Hamilton and Ludwig scales and its inter-variability.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 55 years (both inclusive).
2. Good general health as determined from recent medical history.
3. No previous history of adverse skin conditions, and not under any medication likely to interfere with the results.
4. Patient having androgenic alopecia condition with grade of 1 to 3 (Dermatological assessment)

Exclusion Criteria:

1. Recent hair transplantation or other surgical interventions on the scalp within the past year.
2. Pregnant or breastfeeding women will be excluded due to potential hormonal influences on hair growth.
3. History of cancer treatment involving chemotherapy or radiotherapy to the scalp.
4. Presence of significant dermatological conditions affecting the scalp other than androgenetic alopecia (e.g., psoriasis, severe seborrheic dermatitis).
5. History of major systemic diseases (e.g., uncontrolled diabetes, severe cardiovascular diseases, autoimmune disorders).
6. Any other condition which could warrant exclusion from the study, as per the dermatologist/investigator's discretion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects having Alopecia. (Grade I to III)
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
To establish a standardized methodology that integrates various parameters comprehensively assess and evaluate hair growth and scalp health. | 0n Day 1
To establish a standardized methodology for measurement of hair regrowth from AGA-affected area (bald scalp) and tattoo area. | 0n Day 1
  Evaluated using the standardized area 30 cm from nose tip followed by the CASLite Nova.
To establish a standardized methodology for evaluating number of new hairs from the AGA-affected area (bald scalp) and tattoo area. | 0n Day 1
  Evaluated using the standardized area 30 cm from nose tip followed by the CASLite Nova.
To establish a standardized methodology for evaluation of hair strength through tensile testing | 0n Day 1
  Evaluated using TESTRONIX Instrument.
To establish a standardized methodology for assessment of hair length | 0n Day 1
  Evaluated using the standardized area 15 cm away from the tip of the nose towards scalp vertex.
To establish a standardized methodology for assessment of Global picture of head crown | 0n Day 1
  Evaluated digital photographs of the alopecia at 0° Angle, 45° Angle, 90° Angle.
To establish a standardized methodology for assessment of quantitative scalp keratin assessment. | 0n Day 1
  Evaluated using CASLite Nova Instrument
To establish a standardized methodology for assessment of quantitative hair keratin assessment. | 0n Day 1
  Evaluated using Bradford Assay.
To establish a standardized methodology for quantitative scoring of baldness using the Norwood-Hamilton and Ludwig scales and its inter-observer variability. | 0n Day 1
  Evaluated using certified Dermatologist where type I = Minimal recession of the hairline and type Va indicates Most advanced degree of alopecia

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Maheshvari N Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No